CLINICAL TRIAL: NCT03909503
Title: A Case Series Evaluating a Porcine-derived Collagen Wound Dressing to Treat Chronic Lower Extremity Wounds
Brief Title: A Case Series Evaluating a Collagen Wound Dressing to Treat Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2018-DIV71-029
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Porcine-derived collagen wound dressing (Experimental): The dressing is a sheet of collagen composed of type I collagen derived from porcine peritoneal membrane. The dressing also contains additional components from the procine extracellular matrix. The dressing is a currently marketed, cleared device in the United States indicated for the management of full- and partial-thickness wounds, including: pressure ulcers, diabetic ulcers, venous ulcers, and several other wound types.
  Interventions: Device: Porcine-derived collagen wound dressing

INTERVENTIONS:
Device: Porcine-derived collagen wound dressing — Patients who meet the inclusion criteria will be treated with porcine-derived collagen dressings. The dressing will be used in accordance with its label. After cleansing the wound, the dressing will be placed on the wound. Appropriate primary and secondary dressings will be placed over the intervention product. Patients will visit the clinic once per week to have their dressings re-applied. Wound evaluations will take place once per week with the intervention lasting up to twelve weeks. Concomitant standard of care such as compression for venous ulcers will be provided according to individual patient needs.

SUMMARY:
Chronic wounds are a source of significant morbidity and escalated healthcare costs. The wound care professional has a myriad of modern wound dressings to choose from, each of which has benefits and drawbacks. An understanding of how a given dressing performs in healing a particular wound is crucial in order to determine a clinical mapping of wound dressings to wound types; such a categorization would lead to more efficient clinical decision making and better patient outcomes. This case series will evaluate the ability of a porcine-derived collagen dressing to improve healing of chronic lower-extremity wounds.

ELIGIBILITY:
Inclusion Criteria:

* Has at least one of the following types of wounds below the knee: diabetic ulcer, pressure ulcer, venous ulcer, ulcer of mixed-vascular origin, traumatic wound, post-surgical wound
* Wound has been present for at least four weeks
* Wound is free of necrotic tissue or it is possible for necrotic tissue to be removed by typical debridement practices prior to or during treatment phase
* Wound has not healed after using at least one other type of advanced wound care treatment
* Wound size is between 1 and 100 cm2
* Patient has adequate circulation, as demonstrated by biphasic or triphasic Doppler waveform, measured within three months prior to study enrollment. If monophasic on exam, then non-invasive tests must display Ankle Brachial Index greater than 0.8 and no worse than mild disease on segmental pressures.
* Wound is free of infection and absence of osteomyelitis.

Exclusion Criteria:

* Pregnant, planning to become pregnant during the study timeframe, or breast feeding
* Has a known allergy to porcine products
* Has an allergy or sensitivity to any type of collagen
* Unable or unwilling to receive porcine collagen
* Wound is infected or there is presence of osteomyelitis
* Inability, in the opinion of the Investigator to follow protocol requirements, attend follow up visits in a timely manner, or otherwise comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in wound size over a twelve week period | Baseline to 84 days

SECONDARY OUTCOMES:
Bates-Jensen Wound Assessment Tool score | Baseline to 84 days
  The Bates-Jensen Wound Assessment tool score will be used to assess the wound's status throughout the study. The wound size score ranges from 0 to 5. The wound depth score ranges from 0 to 5. The wound edge score ranges from 0 to 5. The wound undermining score ranges from 0 to 5. The necrotic tissue type score ranges from 1 to 5. The necrotic tissue amount ranges from 1 to 5. The exudate type score ranges from 1 to 5. The exudate amount score ranges from 1 to 5. The skin color surrounding wound score ranges from 1 to 5. The peripheral tissue edema score ranges from 1 to 5. The peripheral tissue induration score score ranges from 1 to 5. The granulation tissue score ranges from 1 to 5. The epithelialization score ranges from 1 to 5. The total score from these sub-scores added together is used as the total BWAT score. For all sub-score values, a value of 0 or 1 is a better outcome. A score of 1 indicates the healthiest and 5 indicates the unhealthiest attribute for each characteristic.
Change in reported pain level: verbal numeric pain rating scale | Baseline to 84 days
  The pain will be recorded using a verbal numeric pain rating scale from 0 to 10. A score of 0 indicates no pain and a score of 10 indicates the highest rated pain.

IPD SHARING:
Plan to Share IPD: No